CLINICAL TRIAL: NCT06752746
Title: A Phase Ib, Multicenter, Randomized, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of 9MW3011 in Patients With Polycythemia Vera
Brief Title: A Study of Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of 9MW3011 in Patients With Polycythemia Vera
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9MW3011-C03
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Open-label 9MW3011 Dose1 (Experimental): Drug: 9MW3011 9MW3011 for multiple dose via intravenous infusion
  Interventions: Drug: 9MW3011
- Experimental: Open-label 9MW3011 Dose2 (Experimental): Drug: 9MW3011 9MW3011 for multiple dose via intravenous infusion
  Interventions: Drug: 9MW3011
- Experimental: Open-label 9MW3011 Dose3 (Experimental): Drug: 9MW3011 9MW3011 for multiple dose via intravenous infusion
  Interventions: Drug: 9MW3011

INTERVENTIONS:
Drug: 9MW3011 — Multiple dose

SUMMARY:
The goal of this clinical trial is to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of 9MW3011 in Chinese patients with Polycythemia Vera（PV）.

DETAILED DESCRIPTION:
The multiple dose fo the starting dose cohorts will comprise 3 dose cohorts of 8 PV subjects each.In each cohort, subjects will receive 9MW3011 via intravenous infusion.A decision on whether to proceed with case expansion and dose escalation will be based on the safety and PK-PD data.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years or older at the time of screening.
2. A confirmed diagnosis of PV according to the revised 2016 World Health Organization criteria and are resistant to or intolerant of hydroxyurea or Interferon alpha.
3. Have a treatment history for PV with resistance or intolerance to hydroxyurea or Interferon alpha.
4. Subjects receiving hydroxyurea, Interferon alpha, or ruxolitinib must complete a washout period before administration of the investigational drug.
5. Must agree to adhere to appropriate contraception requirements during the study period.
6. All female subjects with fertility capacity tested negative for blood pregnancy.
7. Voluntarily participate in clinical trials and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

1. The spleen is palpable at least 5 centimeters below the left costal margin upon palpation at baseline.
2. Heart failure, unstable angina pectoris, myocardial infarction, and other thrombotic diseases within the 6 months prior to screening.
3. Abnormal QTc interval of electrocardiogram within the 6 months prior to screening.
4. Uncontrolled hypertension prior to screening.
5. Any non-PV myeloproliferative neoplasms (MPN).
6. Blast cells and blast granulocytes in the peripheral blood within the 3 months prior to screening.
7. Hematological indicators do not meet the requirements at the time of screening.
8. Known positive for active hepatitis B, hepatitis C, syphilis or human immunodeficiency virus (HIV) infection.
9. History of invasive malignancies within the last 5 years.
10. Severe infection or uncontrolled active infection.
11. Other hematological and lymphatic system diseases or any diseases causing hemolysis or erythrocyte instability.
12. Other systemic diseases or a family history of systemic diseases, may affect the subject's safety or any other diseases and physiological conditions that may affect the results of the study, judged by the investigator.
13. Specific history of allergies.
14. Subjects who have used monoclonal antibodies within the 6 months prior to screening.
15. Patients who have received vaccinations within 6 weeks prior to screening.
16. Subjects who have received other antitumor therapeutic drugs for PV prior to screening.
17. Chronic diseases requiring treatment with systemic glucocorticoids or other immunosuppressants.
18. History of drug abuse or illicit drug use within 3 months prior to screening.
19. Participation in other clinical trials within 3 months prior to screening.
20. Planned elective surgery during the study.
21. History of surgery within 3 months prior to screening.
22. Intolerable iron deficiency-related symptoms judged by the investigator prior to the first dosing.
23. Pregnant or lactating females; women of reproductive age who are not using effective contraception.
24. Individuals directly associated with the research and/or their immediate family members.
25. Other factors which may potentially affect the assessment of the study results by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | Up to 141 or 197 days
  Incidence of adverse events
Vital sign | Up to 141 or 197 days
  Incidence of treatment-emergent clinically abnormal vital signs
Physical examination | Up to 141 or 197 days
  Incidence of treatment-emergent clinically abnormal physical examinations
12-lead electrocardiogram (ECG) | Up to 141 or 197 days
  Incidence of treatment-emergent clinically significant 12-lead electrocardiograms (ECGs)
Laboratory test result | Up to 141 or 197 days
  Incidence of treatment-emergent clinically significant laboratory test results

SECONDARY OUTCOMES:
Cmax | Day 1 to Day 141 or 197
  Plasma maximum measured drug concentration
Tmax | Day 1 to Day 141 or 197
  Time of maximum concentration
AUC0-τ | Day 1 to Day 141 or 197
  Area under the plasma concentration-time curve during a dosage interval（τ）
AUC0-t | Day 1 to Day 141 or 197
  Area under the concentration-time curve from dosing to the last measurable time point
AUC0-∞ | Day 1 to Day 141 or 197
  Area under the concentration-time curve from dosing to infinity
λz | Day 1 to Day 141 or 197
  Terminal elimination rate constant
t1/2z | Day 1 to Day 141 or 197
  The terminal elimination half-life
MRT | Day 1 to Day 141 or 197
  Mean residence time
Vss | Day 1 to Day 141 or 197
  Volume of Distribution at Steady State
CLss | Day 1 to Day 141 or 197
  Steady-state clearance
DF | Day 1 to Day 141 or 197
  Fluctuation percentage
Ctrough | Day 1 to Day 141 or 197
  Trough Concentration
Rac(AUC) | Day 1 to Day 141 or 197
  Accumulation ratio calculated from the AUCτ,ss and AUCτ after single dosing
Rac(cmax) | Day 1 to Day 141 or 197
  Accumulation ratio calculated from the Cmax,ss and Cmax after single dosing
Hepcidin | Day 1 to Day 141 or 197
  Change from baseline in hepcidin levels
Serum iron | Day 1 to Day 141 or 197
  Change from baseline in serum iron levels
Transferrin saturation (TSAT) | Day 1 to Day 141 or 197
  Change from baseline in transferrin saturation (TSAT) levels
Anti-drug antibodies(ADA) | Day 1 to Day 141 or 197
  The incidence of ADA
Hematocrit (HCT) | Day1 to Day 141 or 197
  Change from baseline in HCT levels
Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score（MPN-SAF TSS） | Day 1 to Day 141 or 197
  Change from baseline in MPN-SAF TSS score

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Affiliated Cancer Hospital of Zhengzhou University and Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang